CLINICAL TRIAL: NCT02549638
Title: Identification of Prognostic Biomarkers for Progression of Invasive Squamous Cell Carcinoma
Status: Terminated | Type: Observational
Why Stopped: Lack of funding, slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, PI, Mayo Clinic
Other Study IDs: 15-000548
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Squamous Cell; Carcinoma, Squamous; Squamous Cell Carcinoma; Lung Neoplasms; Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms
MeSH Terms: conditions — Carcinoma, Squamous Cell; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 bronchoscopic biopsies, 10ml blood and one tumor and adjacent normal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tissue Collection: We plan to prospectively collect 5 bronchoscopic biopsies, 3ml blood and one tumor and adjacent normal samples from 200 qualified patients who meet the study criteria. If a patient has already had a bronchoscopy and has samples available that were previously collected and stored for research at the Mayo Clinic we will use those samples.
  Interventions: Genetic: DNA Extraction

INTERVENTIONS:
Genetic: DNA Extraction — We will then extract DNA from tissue sections and blood and use a custom targeted sequencing panel of 23 cancer driver genes with significant mutations in squamous cell carcinoma that we have developed to find the prognostic biomarkers. The DNA will be used in a PCR reaction to generate amplicons for library preparation using Illumina Nextera XT library preparation protocol and targeted sequencing on the Illumina Hiseq sequencer. The reads will be aligned to the HG19 using BWA aligner and variant detection performed with Agilent SureCall and GATK analytic tools.

SUMMARY:
The study will utilize both retrospective and prospective data collection from patients that already had a bronchoscopy and lung resection or will have a bronchoscopy and lung resection for squamous cell carcinoma. The investigators plan to prospectively collect 5 bronchoscopic biopsies, 10ml blood and one tumor and adjacent normal samples from 200 qualified patients who meet the study criteria.

DETAILED DESCRIPTION:
The study will utilize both retrospective and prospective data collection from patients that have already had a bronchoscopy and lung resection or will have a bronchoscopy and lung resection for squamous cell carcinoma. The investigators plan to prospectively collect 5 bronchoscopic biopsies, 10ml blood and one tumor and adjacent normal samples from 200 qualified patients who meet the study criteria. If a patient has already had a bronchoscopy and has consented to have samples stored for research at the Mayo Clinic Rochester we will access them for the research study if available. Otherwise, if the patient has already had surgery and tissue has not been stored for research the investigators will consent patients to use their clinical specimens for the research study. The investigators will then extract DNA from tissue sections and blood and use a custom targeted sequencing panel of 23 cancer driver genes with significant mutations in squamous cell carcinoma that they have developed to find the prognostic biomarkers. The DNA will be used in a PCR reaction to generate amplicons for library preparation using Illumina Nextera XT library preparation protocol and targeted sequencing on the Illumina Hiseq sequencer. The reads will be aligned to the HG19 using BWA aligner and variant detection performed with Agilent SureCall and GATK analytic tools.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected squamous cell carcinoma of the lung
* able to provide consent
* could have already had a bronchoscopy or surgical resection with tissue saved at the Mayo Clinic Rochester
* will be undergoing a bronchoscopy and having a surgical resection at the Mayo Clinic Rochester

Exclusion Criteria:

* unable to provide consent
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Thoracic Surgery Patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Number and types of recurrent genomic alterations evaluated by a custom targeted sequencing panel. | 2 years
  The aim of this study is to identify and characterized recurrent genomic alteration found in invasive squamous cell carcinoma that are present in the precursor airway epithelial tissues but absent in normal tissues examined from samples taken during a lung procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials